CLINICAL TRIAL: NCT01674127
Title: Effect of Methyldopa on Uterine Artery Diameter in Pregnant Women With Mild Preeclampsia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mojtaba Akbari, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 390306
Record Dates: First submitted 2012-08-24; First posted 2012-08-28 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-08

CONDITIONS: Pregnant Women With Mild Preeclampsia
MeSH Terms: interventions — Methyldopa

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Methyldopa (Experimental): In case group, 25 patients, under treatment, using Methyldopa for 7 days, received 500 mgs of Methyldopa in its oral form per day and in control group, participants received placebo for 7 days.
  Interventions: Drug: Methyldopa
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methyldopa
  Arms: Methyldopa
Drug: Placebo
  Arms: placebo

SUMMARY:
The present study examined the effects of Methyldopa on uterine artery diameter, uterine artery blood flow, umbilical artery and fetal middle-cerebral artery in patients with Preeclampsia, using Doppler ultrasound.

ELIGIBILITY:
They met the inclusion criteria, If they had over 25 weeks of gestational age, no history of chronic hypertension, no diabetes mellitus, no chronic systemic diseases, no collagen vascular diseases and antiphospholipid syndromes, no use of antihypertensive drugs and BMI higher than 19 and lower than 30 (kg/m2).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-08; Primary Completion 2012-02 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Doppler indices | 7 days
  In case group, 25 patients, under treatment, using Methyldopa for 7 days, received 500 mgs of Methyldopa in its oral form per day and in control group, participants received placebo for 7 days.Before and after drug use, Doppler ultrasound test was done by a radiology specialist not informed of patients grouping. Also, pulsatility index, resistance index, systolic/diastolic blood flow ratios of uterine artery, umbilical artery and middle-cerebral artery were evaluated. Registered for all patients, age, BMI, gestational week and the number of pregnancies were among other examined variables.
  Doppler indices of examined arteries in studied groups were evaluated by color Doppler ultrasound of model "Hitachi 3/6 MHz".